CLINICAL TRIAL: NCT00477087
Title: Phase II Study of Granulocyte-Macrophage Colony Stimulating Factor Plus Mitoxantrone for the Treatment of Hormone Refractory Prostate Cancer
Brief Title: Phase II GM-CSF Plus Mitoxantrone in Hormone Refractory Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Stanford University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Sandy Srinivas, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-04738; 96817 (Other: Stanford University alternate IRB Number); PROS0017 (Other: OnCore Number)
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Mitoxantrone; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GM-CSF Plus Mitoxantrone (Experimental): GM-CSF at 250 micrograms/ m² / day subcutaneously 3 x week for 3 weeks. Participants will also receive mitoxantrone 14 mg/m² on Day 1 of each cycle. Each cycle of therapy consists 21 days.
  Interventions: Drug: Mitoxantrone; Drug: GM-CSF

INTERVENTIONS:
Drug: Mitoxantrone — Mitoxantrone is an anti-cancer chemotherapy drug that is classified as an antitumor antibiotic.
  Other Names: Novantrone
Drug: GM-CSF — GM-CSF is a biologic response modifier, classified as a colony stimulating factor.
  Other Names: Sargramostim; Leukine; Granulocyte-Macrophage Colony Stimulating Factor

SUMMARY:
The purpose of this study is to evaluate the effect of the combination of mitoxantrone and granulocyte-macrophage colony stimulating factor (GM-CSF) on progression-free survival (PFS) and overall survival (OS), in patients with hormone-refractory prostate cancer.

DETAILED DESCRIPTION:
This trial evaluates if the addition of GM-CSF to standard-of-care therapy after 1st-line docetaxel improves tumor control and survival. Because the 2 drugs have completely different mechanisms of action as well as non-overlapping metabolism, clinically significant drug-drug interactions are not anticipated, and therefore both drugs will be given at standard (approved) doses.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age ≥ 18 years
* Histologically-confirmed adenocarcinoma of the prostate
* Hormone-refractory prostate cancer
* Failed 1st-line docetaxel-containing regimen
* No prior immunotherapy including:

  * Vaccines
  * GM-CSF
* Minimum prostate-specific antigen (PSA) > 5 mg/dL and rising according to the PSA Consensus Criteria
* Karnofsky Performance Status (KPS) > 60%
* Eastern Cooperative Oncology Group (ECOG) Performance Status < 3
* Life expectancy > 6 months

Exclusion Criteria:

* Concomitant hormonal therapy other than luteinizing hormone-releasing hormone (LHRH) agonist
* Use of herbal products known to decrease PSA levels
* Use of supplements or complementary medicines, except for:

  * Conventional multivitamin supplements
  * Selenium
  * Lycopene
  * Soy supplements
  * Vitamin E
* Initiation of bisphosphonates within one month prior to enrollment or throughout the study
* Any prior radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment
* Major surgery or radiation therapy completed < 4 weeks prior to enrollment
* Any concomitant second malignancy other than non-melanoma skin cancer
* Any concomitant serious infection
* Any nonmalignant medical illness
* Absolute neutrophil count (ANC) < 1,500/µL
* Platelet count < 100,000 µL
* Hemoglobin < 8 mg/dL
* Total bilirubin greater than 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN if no demonstrable liver metastases, or greater than 5.0 x ULN in presence of liver metastases
* Ejection fraction < 50% as measured by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
* Noncompliance with study procedures

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — males (prostate cancer)
Enrollment: 10 (Actual)
Dates: Start 2006-07; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GM-CSF Plus Mitoxantrone
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GM-CSF Plus Mitoxantrone
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Assessed as the time from the 1st dose of study drug to death or disease progression (increase >25% over baseline PSA on 2 consecutive measurements 2 weeks apart, need for palliative therapy, formation/progression of new bone lesions, or decline of >20% KPS)
Time Frame: 18 months
Measure: Median (Full Range); unit: weeks
Arm/Group | GM-CSF Plus Mitoxantrone
Number analyzed (Participants) | 10
weeks | 7.5 [3 to 40]

2. Secondary Outcome: Number of Participants With > 50% Decrease in Prostate-specific Antigen Levels (PSA Response)
Description: Defined as the first evidence of a total serum PSA decline of > 50% from baseline, maintained for at least 28 days, and confirmed with 2 consecutive measurements taken 2 weeks apart.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | GM-CSF Plus Mitoxantrone
Number analyzed (Participants) | 10
Participants | 3

3. Secondary Outcome: Overall Survival (OS)
Description: Assessed as the time from the 1st dose of study drug to death.
Time Frame: 18 months
Measure: Median (Full Range); unit: Months
Arm/Group | GM-CSF Plus Mitoxantrone
Number analyzed (Participants) | 10
Months | 7.8 [3 to 12.6]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | GM-CSF Plus Mitoxantrone
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF Plus Mitoxantrone (N=10)
Hematuria (Blood and lymphatic system disorders) | 1 (1)
Pancytopenic (Blood and lymphatic system disorders) | 1 (1)
Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Death due to progressive disease
Acute renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GM-CSF Plus Mitoxantrone (N=10)
Fatigue (General disorders) | 6 (6)
Diarrhea (General disorders) | 1 (1)
Dizziness (Eye disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Dyspnea (Infections and infestations) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Night sweats (Nervous system disorders) | 3 (3)
Weight gain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes